CLINICAL TRIAL: NCT02636985
Title: Transthoracic Ultrasound Elastography in Pulmonary Lesions and Diseases
Brief Title: Application of Ultrasonic Elastography in Lung Lesions
Status: Completed | Type: Observational
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 201503075RINC
Record Dates: First submitted 2015-11-24; First posted 2015-12-22 (Estimated); Last update posted 2015-12-22 (Estimated); Status verified 2015-12

CONDITIONS: Elastography

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Elastography is an imaging of tissue elasticity or stiffness and is currently emerging as a mainstream tool for ultrasound-based diagnosis. This compressibility property of materials, mathematically expressed as the change in tissue displacement as a function of its distance from the compressing device, is known as strain and is the parameter that is imaged in an elastogram.

Elastography has currently shown promising result in differentiating viscoelastic nature of various organs, which is a consequence of certain underlying diseases.

At present, there are limited literatures revealing the application and feasibility of ultrasonic elastography in lung lesions. This is essentially important as it may serve as an adjuvant to B-mode ultrasound. The investigators aimed at exploring the application and feasibility of ultrasonic elastography on lung lesions.

DETAILED DESCRIPTION:
Patients performed conventional B-mode ultrasound, subsequently followed by ultrasound elastography. The strain ration was measured and was compared between necrosis, atelectasis, consolidation and tumor.

ELIGIBILITY:
A. Inclusion Criteria:

Patients with radiographic findings of:

1. consolidation
2. obstructive pneumonitis
3. tumors

B. Exclusion Criteria:

1. Patients with poor acoustic window
2. Unable to hold breathing
3. Not cooperative
4. Presence of pleural effusion

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with radiographic findings of consolidation, obstructive pneumonitis or tumors, detected on chest computed tomography (CT), who received ultrasound study with or without ultrasound-guided biopsy for tissue proof and UE, from December 2011 to March 2013.
Sampling Method: Probability Sample
Enrollment: 45 (Actual)
Dates: Start 2011-12; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
Comparison of strain ratio between necrosis, atelectasis, consolidation and tumor | Up to 15 months
  The strain ratio was measured under ultrasonic elastography. At least three measurements were performed each time and we average all the measurements as the final strain ratio. Independent t test was used for comparison.

CONTACTS AND LOCATIONS:
Overall Officials: Hao-Chien Wang, MD, PhD, Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taipei City, Taiwan

REFERENCES:
- [Derived] Lim CK, Chung CL, Lin YT, Chang CH, Lai YC, Wang HC, Yu CJ. Transthoracic Ultrasound Elastography in Pulmonary Lesions and Diseases. Ultrasound Med Biol. 2017 Jan;43(1):145-152. doi: 10.1016/j.ultrasmedbio.2016.08.028. Epub 2016 Oct 12. PMID 27743728